CLINICAL TRIAL: NCT05708495
Title: Efficacy of Adding Posterior Ilium Mobilization With Movement to Treatment of Patellofemoral Pain Syndrome
Brief Title: Ilium Mobilization in Patellofemoral Pain Syndrome Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Labib Mousa Labib Ghali, Assistant Lecturer Of Orthopedic Physical Therapy, Faculty Of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ilium mobilization
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-09

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; strength; stretch; mobilization; ilium; innominate
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: strengthening and stretching exercises
- Study group (Experimental)
  Interventions: Other: posterior ilium mobilization; Other: strengthening and stretching exercises

INTERVENTIONS:
Other: posterior ilium mobilization — the therapist will mobilize the innominate on the affected side posteriorly
  Arms: Study group
Other: strengthening and stretching exercises — the participants will receive strengthening exercises on the hip and knee joint beside that they will receive stretching exercises

SUMMARY:
Aim of the study is to investigate the effect of adding posterior ilium mobilization on knee pain, knee function, anterior pelvic tilt, dynamic knee valgus, muscle strength of extensors, abductors and external rotators of hip and knee extensors in patients with patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the subjects between 18-35 years.
2. BMI will be ≤ 29.5
3. Anterior or retro patellar knee pain for at least 6 weeks duration.
4. Foot posture index score from +6 to +12.
5. Anterior pelvic tilt angle more than 8 degree.
6. Pain elicited at least by two of the following four tests; (i) Isometric muscle contraction with slight bent knee,(ii) palpation of the patellofemoral joint line, (iii) patellar compression against the femoral bone (iv) active resisted knee extension.
7. Pain intensity more than 3 at ANPS and provoked by at least two of the following activities: running, walking, hopping, squatting, stair negotiation, kneeling, or prolonged sitting.

Exclusion Criteria:

1. Meniscal or other intraarticular pathologic conditions; cruciate or collateral ligament involvement.
2. A history of traumatic patellar subluxation or dislocation.
3. Previous surgery in the knee, ankle and hip joints.
4. Knee, ankle and hip joints osteoarthritis.
5. Taking non-steroidal anti-inflammatory drugs or corticosteroids within 24 h before the test.
6. History of brain injury or vestibular disorder within the last 6 months.
7. Pregnant female.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in pain | It will be assessed at baseline and after 4 weeks
  Arabic Numeric pain rating scale will be used to assess pain changes during walking, hopping, squatting, stair negotiation, kneeling, or prolonged sitting.
  This scale measures pain severity on a scale of 0 to 10 points, with 0 representing no pain and 10 signifying the most severe pain possible.
Changes in knee functional disability | It will be assessed at baseline and after 4 weeks
  The Arabic version of Anterior knee pain scale will be used to assess the knee functional disability.
  It is a self-administered, weighted questionnaire that analyzes 13 items, including pain and function, with a maximum score of 100 points and minimum score of 0 points. Higher scores indicate greater lower extremity function. It documents responses to six activities linked with anterior knee pain (walking, running, jumping, climbing stairs, squatting, and sitting for prolonged periods with knee bent).

SECONDARY OUTCOMES:
Changes in hip abductors strength | It will be assessed at baseline and after 4 weeks
  Handheld dynamometer will be used to assess changes in muscle strength
Changes in hip extensors strength | It will be assessed at baseline and after 4 weeks
  Handheld dynamometer will be used to assess changes in muscle strength
Changes in hip external rotators strength | It will be assessed at baseline and after 4 weeks
  Handheld dynamometer will be used to assess changes in muscle strength
Changes in knee extensors strength | It will be assessed at baseline and after 4 weeks
  Handheld dynamometer will be used to assess changes in muscle strength
Changes in dynamic knee valgus | It will be assessed at baseline and after 4 weeks
  Cell phone Camera, tripod device and Kinovea Computer Program (KCP) will be used to assess knee frontal plane projection angle to detect changes in knee valgus during step down test
Changes in pelvic tilt angle | It will be assessed at baseline and after 4 weeks
  Palpation Meter (PALM) will be used to assess changes in pelvic tilt angle

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt